CLINICAL TRIAL: NCT04684108
Title: A Phase 1 Study of SG301 in Subjects With Hematological Malignancies
Brief Title: SG301 Safety Study in Subjects With Relapsed or Refractory Multiple Myeloma and Other Hematological Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Sumgen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSG-301-101
Record Dates: First submitted 2020-12-10; First posted 2020-12-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Relapsed or Refractory Multiple Myeloma; Hematological Malignancy
MeSH Terms: conditions — Recurrence; Multiple Myeloma; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SG301 (Experimental): SG301 monotherapy intravenous (IV) infusion
  Interventions: Drug: SG301

INTERVENTIONS:
Drug: SG301 — Phase 1a will use an accelerated titration and 3+3 design with 9 dose cohorts: 0.005 mg/kg, 0.05 mg/kg,0.5 mg/kg, 1 mg/kg, 2 mg/kg, 4 mg/kg, 8 mg/kg, 12 mg/kg and 16 mg/kg by IV infusion. Accelerated titration (i.e., 1 patient each) will be applied to the first 3 cohorts.

SUMMARY:
This is a Phase 1a/1b Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SG301 in Patients with Relapsed or Refractory Multiple Myeloma and Other Hematological Malignancies

DETAILED DESCRIPTION:
After a screening period of up to 28 days for each study phase, qualified patients will be enrolled to receive their assigned dose of SG301, administered weekly for the first 2 cycles and every 2 weeks thereafter, until disease progression or intolerable toxicity, starting of a new anticancer treatment, withdrawal of consent, lost to follow up, death, or end of the study, whichever occurs first.

The study consists of a dose escalation phase (Phase 1a) and a dose expansion phase (Phase 1b) in subjects with relapsed or refractory multiple myeloma and other hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form (ICF).
2. Age ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1 or 2.
4. Expected survival time of ≥3 months.
5. Patients with histologically or cytologically confirmed hematological malignancies who are relapsed or refractory to or intolerant of standard therapies.

   For patients with multiple myeloma: should be relapsed or refractory multiple myeloma with measurable disease
6. Adequate organ function
7. Toxicity caused by prior anti-tumor therapy recovered to Grade 0 to 1 (CTCAE 5.0), except for alopecia, controlled Grade ≤2 sensory neuropathy, lymphocytopenia, and endocrine disorders.
8. Female patients of childbearing potential and male patients whose female partners are of childbearing potential need to use at least one approved contraceptive (e.g., intrauterine device, pill, or condom) during study treatment and for at least 6 months (180 days) after the last dose; female patients of childbearing potential must have a negative blood human chorionic gonadotropin (HCG) test during screening period and must not be lactating.

Exclusion Criteria:

Patient Exclusion Criteria:

1. Presence of central nervous system metastatic lesions.
2. uncontrolled cardiac disease requiring treatment, congestive heart failure NYHA III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 6 months.
3. Active infection requiring antimicrobial therapy within 2 weeks prior to study drug administration.
4. Patients with active viral hepatitis (any etiology) are excluded.
5. Anticancer therapy within 5 half-lives or 2 weeks (whichever is longer)
6. Primary refractory to previous anti-CD38 therapy.
7. Major surgery within 4 weeks prior to study entry.
8. Prior or concurrent malignancy within 2 years prior to entry, other than adequately controlled skin basal cell carcinoma, cervical carcinoma in situ, breast carcinoma in situ, skin squamous cell carcinoma.
9. Any other condition that, in the opinion of the Investigator, may lead to inappropriate participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of one year
  Number and percentage of AE which is calculated by worst CTCAE grade by CTCAE 5.0
MTD/MAD/ RP2D | Through study completion, an average of one year
  To determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) for intravenous (IV) administration of SG301 in patients with relapsed or refractory multiple myeloma and other hematological malignancies; To preliminarily determine the recommended Phase 2 dose (RP2D) of SG301 given intravenously in patients with relapsed or refractory multiple myeloma and other hematological malignancies.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): AUC | Through study completion, an average of one year
  The area under the curve (AUC) of serum concentration of the drug after the administration
Pharmacokinetics (PK): Cmax | Through study completion, an average of one year
  Maximum concentration(Cmax) of the drug after administration
Pharmacokinetics (PK): limination half-life (T 1/2) | Through study completion, an average of one year
  Descripition: limination half-life (T 1/2) of the drug after administration
receptor occupancy (RO) | Through study completion, an average of one year
  receptor occupancy (RO) of CD38 on the surface of peripheral blood cells
Immunogenicity endpoints | Through study completion, an average of one year
  levels of anti-drug antibodies (ADAs) and neutralizing antibodies (tested in ADA-positive samples only).
Efficacy endpoints | Through study completion, an average of one year
  objective response rate (ORR)

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Affiliated Beijing Chaoyang Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Beijing Jishuitan Hostipal, Beijing, Beijing Municipality
  - Shenzhen Second People's Hospital, Shenzhen, Guangzhou
  - The Fourth Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan University Central South Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Wuxi Central Hospital, Wuxi, Jiangsu
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanxi Norman Bethune Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No